CLINICAL TRIAL: NCT04419961
Title: Sexual Dysfunction and an Educational Program to Improve the Quality of Sexual Function in Vietnamese Pregnant Women in First Trimester
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Hospital of Obstetrics and Gynecology (Other)
Responsible Party: Principal Investigator, PHAN CHI PHAN, Principal Investigator, National Hospital of Obstetrics and Gynecology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PSD20
Record Dates: First submitted 2020-06-03; First posted 2020-06-09 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Female Sexual Dysfunction
Keywords: sexual dysfunction; pregnant women; education
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Routine care.
- Intervention (Experimental): Routine care plus participation in an educational program including a group discussion and a booklet.
  Interventions: Behavioral: Educational program

INTERVENTIONS:
Behavioral: Educational program — The educational program includes a group discussion and a booklet.
  The group discussion lasts for 90 minutes, discussing importance of sexual activity during pregnancy, improving sexual experience during pregnancy, physical and mental changes of pregnant women, and measures to cope with discomfort, anxiety, fear and other issues. It includes a 30-minutes presentation, followed by 1-hour discussion.
  The booklet is a color-printed A5-size booklet containing in-depth information of the content given during the discussion. Each participant can only receive one copy of the booklet, and the booklet is not given to the control participants.
  Arms: Intervention

SUMMARY:
Sexual dysfunction is common in pregnant women (46.6%, 34.4%, and 73.3% in women in the first, second, and third trimester worldwide, respectively). These dysfunctions can persist after childbirth, affecting quality of life, marriage satisfaction, and family happiness. In Vietnam, a country heavily influenced by the Eastern traditions, sexual activity is considered private and only shared between husband and wife. Many women have wrong beliefs that having sexual intercouse during pregnancy will affect the safety of the fetus, and thus, are reluctant to engage in sexual activity with their husband. Interventions have been developed to improve the quality of sexual function in pregnant women.

In Vietnam, data of sexual dysfunction in pregnant women are somewhat limited, and there have been no programs to improve the sexual function for this population. Therefore, the study team plans to develop an educational program with aim to improve the quality of sexual function in Vietnamese pregnant women. This study aims to investigate the prevalence and associated factors of sexual dysfunction in first-trimester pregnant women and evaluate the effectiveness of the educational program.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women whose gestational age is less than or equal to 12 weeks.
* Currently living with husband/partner.
* No signs and symptoms of first trimester complications (eg, threated abortion).

Exclusion Criteria:

* Getting pregnant from in vitro fertilization or having a history of preterm birth.
* Having serious health conditions that require abortion.
* Illiterate, or having mental illness or incapacity.
* Having a fetus diagnosed with anomalies.
* Does not agree to participate.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of sexual dysfunction in pregnant women | Baseline
  Sexual function is evaluated using the Female Sexual Function Index (FSFI). The FSFI includes 19 questions covering six domains: desire, arousal, lubrication, orgasm, satisfaction, and pain. Questions ask about participant's sexual experience during the past four weeks, rating the degree/frequency of their experience on a scale from "not at all" or "never" to "very" or "always". Four questions score 1-5 and fifteen score 0-5. Then, the scores of questions in an individual domain are added and the total score is multiplied by the domain factor. Finally, the six domain scores are added to obtain the full scale score. A total FSFI score of <= 26.55 is considered sexual dysfunction.
Change in the FSFI score from baseline to two months | Two months
  Patients are followed up after two months and repeated the FSFI. The difference between the baseline total FSFI score and the two-month total FSFI score is calculated. The mean difference is calculated for the intervention and the control arm.

SECONDARY OUTCOMES:
Change in knowledge and attitude at two months | Two months
  Knowledge and attitude are assessed by asking participants whether they agree or disagree with 24 statements. These statements are developed based on the key messages of the educational program. K/A assessment is repeated at two months. We calculate the proportion of participants who have changes in knowledge and attitude after the educational program.

CONTACTS AND LOCATIONS:
Overall Officials: Thanh C Phan, MD, Principal Investigator — National Hospital of Obstetrics and Gynecology
Locations (1):
- National Hospital of Obstetrics and Gynecology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No